CLINICAL TRIAL: NCT02594202
Title: Care of the Prostate Cancer Patient and Prospective Procurement of Prostate Cancer Tissue
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160010; 16-C-0010
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Prostate Cancer
Keywords: Specimen Collection; Carcinogenesis; Prognostic Biomarkers; Molecular Mechanims; Cell Lines; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Adults (= 18 years of age) with biopsy-proven or suspected prostate cancer

SUMMARY:
Background:

Prostate cancer is the most common noncutaneous cancer among men in the U.S. Researchers want to study blood, tissue, and fluid samples of people with prostate cancer. This will help them understand any changes in cells and genes. These changes might lead to the development and progression of prostate cancer. Researchers think the study could lead to new treatments.

Objective:

To understand the changes in cells and genes that lead to the development and progression of prostate cancer. This could lead to new treatments.

Eligibility:

Men ages 18 and older who have or are suspected to have prostate cancer

Design:

Participants will be screened with physical exam and medical history.

Participants will send tissue blocks of their tumor, if possible. If not, they will provide unstained slides of tumor tissue.

Participants may provide samples of blood, urine, saliva, and prostate secretions.

Participants may have imaging tests. They will lie in a machine that takes pictures of their body. These tests include:

MRI of the prostate

CT of the abdomen and pelvis

Chest x-ray

Participants may need a biopsy or surgery for treatment of their cancer. If so, researchers will collect tissue.

Participants may answer questions about their prostate cancer and quality of life.

Participants may have follow-up visits or other treatments. They may have follow-up phone calls every few months.

DETAILED DESCRIPTION:
Background:

* Prostate carcinoma is the second most common malignancy diagnosed in men. Approximately 1 in 6 men will be diagnosed with prostate cancer in their lifetime.
* Understanding the molecular mechanisms and genomic alterations that cause prostate carcinoma will provide the foundation for the development of novel targeted therapeutic agents for this disease. Since 1982 investigators in the Urologic Oncology Branch have been studying the genetic basis of urologic cancers. The identification of the genes for cancer of the kidney has led to the approval by the FDA of a number of new agents for patients with advanced disease. Similarly, it is our goal to study the cancer biology (genomic, molecular, and cellular biology) of prostate carcinoma in order to develop novel treatment strategies.
* Collection of patient tumor samples allows us to study molecular and biologic pathways and develop novel targeted therapies. Correlation of these samples with radiographical findings and clinical outcomes in patients allows us to predict and understand clinical outcomes and possibly develop predictive and/or prognostic biomarkers.

Objective:

Collect blood, urine, saliva, expressed prostatic secretions, and benign and malignant tissue from patients with known or suspected prostate cancer for the purpose of elucidating the molecular mechanisms of carcinogenesis in prostate cancer and ultimately, identifying novel therapeutic targets.

Eligibility:

- Adults with biopsy-proven or suspected prostate cancer who require diagnostic or therapeutic intervention as part of their diagnosis, standard of care treatment, or followup/surveillance for their neoplasm.

Design:

* Tissue acquisition protocol in which normal and malignant prostate cancer tissues may be obtained at the time of clinically indicated diagnostic and/or therapeutic intervention.
* Blood and urine samples for research will be obtained at baseline and follow-up intervals. Expressed prostatic secretions may be collected at baseline and follow-up intervals. Additionally, saliva may be collected at baseline.
* No investigational or experimental therapy will be given as part of this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults (greater than or equal to 18 years of age) with biopsy-proven or suspected prostate cancer (elevated PSA abnormal digital rectal exam (DRE) abnormal prostate MRI, or family history) who require and are willing to undergo diagnostic or therapeutic intervention as part of their diagnosis, standard of care treatment, or follow-up/surveillance for their neoplasm.
  2. ECOG performance status of 0-2
  3. Must be willing and able to provide informed consent
  4. PSA > or equal to 1.0 ng/ml (for patients aged 30 - 49 years) OR
  5. PSA > or equal to 2.5 ng/ml (for patients 50 years or older) OR
  6. Abnormal DRE (i.e. enlarged, asymmetric, nodular, firm or tender) OR
  7. Abnormal prostate MRI finding OR
  8. Family history of first degree relatives (brother or father) with prostate cancer or first-degree relatives (mother or sister) with breast or ovarian cancer

EXCLUSION CRITERIA:

1. Subjects whose comorbidities would preclude diagnostic or therapeutic intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with biopsy-proven or suspected prostate cancer who require diagnostic or therapeutic intervention as part of their diagnosis, standard of care treatment, or follow-up/surveillance for their neoplasm.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-12-21 (Actual); Primary Completion 2036-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Collect samples for the purpose of studying the molecular mechanisms of carcinogenesis in prostate cancer | Ongoing
  Collection of blood, urine, saliva, expressed prostatic secretions, and benign and malignant tissue

SECONDARY OUTCOMES:
prostate cancer cell lines | ongoing
  Develop stable prostate cancer cell lines from procured tissue when feasible
Natural history of prostate cancer | ongoing
  Collect detailed history, pathologic data, perioperative findings, and treatment data to better characterize the natural and clinical histories of prostate cancer when feasible
Molecular profiling | ongoing
  whole genomic sequence characterizations, identification of specific mutations or single nucleotide polymorphisms (SNPs), comparative genomic hybridization, messenger and microRNA sequencing and expression, RNA Seq, DNA methylation (epigenetics), DNA copy number, and expression profiling

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Merriman KM, Harmon SA, Belue MJ, Yilmaz EC, Blake Z, Lay NS, Phelps TE, Merino MJ, Parnes HL, Law YM, Gurram S, Wood BJ, Choyke PL, Pinto PA, Turkbey B. Comparison of MRI-Based Staging and Pathologic Staging for Predicting Biochemical Recurrence of Prostate Cancer After Radical Prostatectomy. AJR Am J Roentgenol. 2023 Dec;221(6):773-787. doi: 10.2214/AJR.23.29609. Epub 2023 Jul 5. PMID 37404084
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0010.html